CLINICAL TRIAL: NCT06086912
Title: A Single-center, Randomized, Open, Three-period, Three-sequence Crossover Clinical Study to Compare the Bioavailability and Safety of a Single Subcutaneous Injection of HR17031 in Healthy Subjects at Different Sites
Brief Title: A Clinical Study to Compare the Bioavailability of HR17031 in Healthy Subjects at Different Sites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR17031-106
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a single-center, randomized, open-label, three-period, and three-sequence crossover design trial, consisting of three sequences (sequence 1, sequence 2 and sequence 3) and three periods (first period, second period and third period). Each sequence receives a same dose of HR17031 at every period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sequence 1 (Experimental)
  Interventions: Drug: HR17031
- sequence 2 (Experimental)
  Interventions: Drug: HR17031
- sequence 3 (Experimental)
  Interventions: Drug: HR17031

INTERVENTIONS:
Drug: HR17031 — Receive a single dose of HR17031 at every period (First period：abdomen. Second period. upper arm. Third period: thigh).
  Arms: sequence 1
Drug: HR17031 — Receive a single dose of HR17031 at every period (First period：upper arm. Second period: thigh. Third period: abdomen).
  Arms: sequence 2
Drug: HR17031 — Receive a single dose of HR17031 at every period (First period：thigh. Second period: abdomen. Third period: upper arm).
  Arms: sequence 3

SUMMARY:
The purpose of this study is to evaluate the bioavailability and safety of HR17031 injection in healthy subjects at different sites.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent form before related activities of the experiment and understanding of the procedures and methods of the experiment, willing to strictly follow the clinical trial protocol to complete the experiment.
2. Both men and women are eligible, aged 18 to 55 years old (inclusive, as determined at the time of signing informed consent form).
3. Body mass index (BMI) is between 18 and 27 kg/m2 (inclusive), with male weight ≥ 50 kg and female weight ≥ 45 kg.
4. Fasting blood glucose level < 6.1 mmol/L during screening period.

Exclusion Criteria:

-

1. The following laboratory or auxiliary examination abnormalities are present during the screening period:

1. Any abnormal laboratory examination with clinical significance. For laboratory examinations with clinical significance, if there is a clear and reasonable reason, retesting can be performed within one week and the retest results used to determine whether the subject meets the criteria;
2. Abnormalities on 12-lead electrocardiogram (ECG) with clinical significance;
3. Positive for hepatitis B surface antigen (HBsAg), positive for hepatitis C antibody (anti-HCV) (or diagnosed as active hepatitis), or positive for syphilis antibody;
4. Positive for human immunodeficiency virus (HIV) serological test.

2. The following diseases or medical history are present:

1. History of hypertension, or systolic blood pressure outside the range of 90-140 mmHg or diastolic blood pressure outside the range of 60-90 mmHg during screening, and judged to have clinical significance by the investigator;
2. Having a life-threatening disease within the past 5 years (except for basal cell carcinoma or squamous cell carcinoma of the skin);
3. Having a severe systemic infection within the past 1 month;
4. Having a history of acute or chronic pancreatitis, symptomatic gallbladder disease, or other risk factors for pancreatitis that may be present;
5. Having a relevant history of gastrointestinal disease with persistent nausea and vomiting, including but not limited to: having had gastroparesis within the past 6 months that required treatment, unstable (worsening) or poorly controlled (persistent nausea and vomiting) gastroesophageal reflux disease (GERD), or surgery that affects gastric emptying;
6. Having a personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN2) with a genetic predisposition;
7. Having a history of any clinically significant disease or condition that the investigator believes may affect the trial results, including but not limited to a history of cardiovascular, endocrine, neurological, digestive, urinary, hematological, immunological, metabolic diseases, or existing diseases in these systems.

3. Medications (prescription or over-the-counter), food supplements, vitamins, and Chinese herbal medicines used within 2 weeks before the start of treatment are prohibited. Local application of eye/nose drops and ointments are allowed.

4. The following conditions are prohibited:

1. Known or suspected allergy to any component of the study drug;
2. Participated in any clinical trial of drugs or medical devices within the past 3 months (determined by the signing of informed consent form);
3. Average daily alcohol intake of more than 15 g within the past week (15 g of alcohol is equivalent to 450 mL of beer, 150 mL of wine, or 50 mL of low-alcohol white wine); alcohol consumption or positive results on alcohol breath test within 48 hours before treatment;
4. Smokers (at least 5 cigarettes per day) or non-smokers who smoked within 48 hours before treatment (including the use of nicotine replacement products);
5. Long-term or within 48 hours before treatment consumption of coffee, tea, chocolate, or soft drinks, such as those containing methylxanthines (theophylline, caffeine, or theobromine) such as cola;
6. Engaging in strenuous exercise, such as weightlifting, sprinting, long-distance running, cycling, swimming, or playing soccer, within 48 hours before treatment;
7. Known or suspected history of drug abuse or positive urine drug screening test during screening; unable or unwilling to abstain from smoking, nicotine gum, or transdermal nicotine patch during the trial; unwilling to abstain from alcohol during the trial;
8. Blood donation within the past month; or blood donation of ≥400 mL within the past 3 months or loss of blood of ≥400 mL due to trauma or major surgery within the past 3 months;
9. Participants with mental or language disabilities who are unable to fully understand or participate in the trial process;
10. Participants with poor compliance or poor venous access, or those with a history of fainting;
11. Pregnant or breastfeeding women;
12. Participants with the ability to reproduce who have plans to conceive within 10 weeks after the last dose of the study drug or refuse to use medically approved contraception (contraception methods are listed in Appendix 1).

5. Any other condition judged by the investigator to interfere with the evaluation of the trial results or to be inappropriate for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
After a single subcutaneous injection of HR17031, the PK parameters of plasma Noiiglutide and serum INS068: Area Under the Concentration versus time curve (AUC0-t) | Start of treatment up to Day 26
After a single subcutaneous injection of HR17031, the PK parameters of plasma Noiiglutide and serum INS068: Area Under the Concentration versus time curve (AUC0-∞) | Start of treatment up to Day 26
After a single subcutaneous injection of HR17031, the PK parameters of plasma Noiiglutide and serum INS068: Maximum Concentration (Cmax) | Start of treatment up to Day 26

SECONDARY OUTCOMES:
After a single subcutaneous injection of HR17031, the PK parameters of plasma Noiiglutide and serum INS068: Time to maximum concentration (Tmax) | Start of treatment up to Day 26
After a single subcutaneous injection of HR17031, the PK parameters of plasma Noiiglutide and serum INS068: Apparent terminal half-life (t1/2) | Start of treatment up to Day 26
After a single subcutaneous injection of HR17031, the PK parameters of plasma Noiiglutide and serum INS068: Clearance (CL/F) | Start of treatment up to Day 26
After a single subcutaneous injection of HR17031, the PK parameters of plasma Noiiglutide and serum INS068: Apparent volume of distribution (Vz/F) | Start of treatment up to Day 26
Safety indicators: Adverse events (AE, including Injection site reactions, Hypoglycemia events, etc.), serious adverse events (SAE). | Screening period up to Day 26
Immunogenicity indicators: anti-Noiiglutide antibodies | Start of treatment up to Day 26
Immunogenicity indicators: anti-INS068 antibodies | Start of treatment up to Day 26

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided